CLINICAL TRIAL: NCT03040674
Title: An Observational Outcomes Study for Autologous Cell Therapy Among Patients With COPD and Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Lung Institute (Industry)
Responsible Party: Principal Investigator, Melissa Rubio, PhD, APRN, Principal Investigator, Lung Institute
Other Study IDs: LI002 Cohort A
Record Dates: First submitted 2017-01-28; First posted 2017-02-02 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: COPD; Interstitial Lung Disease
Keywords: Shortness of breath; Breathlessness; Cellular therapy; Platelet rich plasma; Quality of life; Pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Dyspnea | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cell therapy treated: All patients/participants enrolled will undergo cell therapy
  Interventions: Procedure: Cell therapy

INTERVENTIONS:
Procedure: Cell therapy — Each participant will receive cell therapy with stem cells harvested either from peripheral blood or from bone marrow plus peripheral blood; after harvest, cells are processed and returned to the patient via peripheral circulation on the same day

SUMMARY:
The purpose of the Lung Institute is to collect and isolate a patient's own cells and platelet rich plasma (PRP) and deliver the product back to the patient same-day. Lung Institute's treatment is limited to self- funded patients with chronic lung disease - chronic obstructive pulmonary disease (COPD) and interstitial lung disease (ILD). The patient's cells and platelet rich plasma are collected through venous harvesting.

The hypothesized outcomes of Lung Institute therapy are safety and minimization of adverse events, a perceived improvement in the patient's lung condition (to be determined by their ability to be more physically active; walking greater distances with or without oxygen and improved quality of life scales), an improvement in the FEV1 among COPD patients, the ability to reduce their use of oxygen and possibly to stop it., the ability to function well without the use of rescue inhalers, reduction or ceasing of secondary pulmonary infections, reduction in emergency room visits and exacerbations related to their disease.

DETAILED DESCRIPTION:
Through the collection of outcome data, Lung Institute aims to explore and describe the safety and efficacy of autologous cellular therapy for chronic lung disease with dissemination to the public and to the medical community for the advancement of regenerative medicine. The study aims to confirm the safety of autologous cell therapy, explore the effect of autologous cell therapy treatment on pulmonary function, and to describe the anecdotal quality of life changes of patients following treatment using both quantitative and qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients are included in treatment by self-referral and after consultation with a designated patient coordinator, who determines initial eligibility, and then by the nurse practitioner or physician of the Lung Institute who determines final eligibility for treatment. All eligible and thereby traded patients are eligible for the study

Exclusion Criteria:

* Patients who are unable to provide informed consent, pregnant patients, prisoners, non-English speakers, patients with a history of cancer within the past 5 years, patients with active tuberculosis or pneumonia. In addition, patients on prescribed blood thinners, with a history of breast or prostate cancer of any time frame or with a history of osteoporosis are excluded from the bone marrow harvest option.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all patients treated with cell therapy at Lung Institute Dallas.
Sampling Method: Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rubio, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Lung Institute Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinic webpage — http://lunginstitute.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the clinic site in Dallas, Texas. Participants were all diagnosed with either COPD or interstitial lung disease by their personal pulmonologist. Records review by provider including diagnosis, past medical history, medications, labs from within 3 months, lung function test results and the participants' ability to travel to and from the treatment site were assessed prior to approval. This study is IRB approved and each participant signed Informed Consent.
Pre-assignment Details: All participants who started in the study were contacted at least twice at 3- and 6- months post-treatment by phone for quality of life follow-up. Participants were lost to follow-up at each time interval if they did not answer or return the call.
Groups:
- Cell Therapy Treated: All patients/participants enrolled will undergo cell therapy
  Cell therapy: Each participant will receive autologous cellular therapy with cells harvested either from peripheral blood or from bone marrow plus peripheral blood. After harvest, cells are processed using minimal manipulation for platelet-rich plasma/ platelet concentrate (from peripheral blood) and/or mesenchymal stem cells (from bone marrow) and returned to the patient via peripheral circulation on the same day.
Period: Overall Study
Arm/Group | Cell Therapy Treated
Started | 489
Participants Completing 3 Month Survey | 351
Participants Completing 6 Month Survey | 241
Completed (Total number of participants completing the study (6 months post-treatment)) | 241
Not Completed | 248
Not completed — Lost to Follow-up | 225
Not completed — Death | 23

BASELINE CHARACTERISTICS:
Population: 489 participants were assessed at baseline
Groups:
- Cell Therapy Treated: All patients/participants enrolled will undergo cell therapy
  Cell therapy: Each participant will receive cell therapy with cells harvested either from peripheral blood or from bone marrow plus peripheral blood; after harvest, cells are processed and returned to the patient via peripheral circulation on the same day
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 489
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 125
  >=65 years | 364
Age, Continuous [Mean (Full Range); unit: years] | 70.59 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 8
  White | 461
  More than one race | 1
  Unknown or Not Reported | 12
Chronic Lung Disease Diagnosis [Count of Participants; unit: Participants]
  Chronic Obstructive Pulmonary Disease (COPD) | 357
  Interstitial Lung Disease (ILD) | 132

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life (QOL) From Baseline
Description: • Change from baseline in overall perceived quality of life over the course of a 6 month period as measured by the Clinical COPD Questionnaire (CCQ). The CCQ is a 10-item questionnaire scored as 0-6 for each item (0 being never and 6 being all the time with higher scores representing worse quality of life). The total score is 0-60.
  The change from baseline over the course of 6 months using the participant's self-reported responses to the CCQ. Higher total values on the CCQ demonstrate worsening quality of life.
Time Frame: Measurements pre-treatment then at 3 and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 489
score on a scale
  Baseline CCQ Score | 35.35 (10.56)
  CCQ Score 3-Months Post-Treatment | 27.96 (10.84)
  CCQ Score 6 Months Post-Treatment | 26.87 (10.84)

2. Primary Outcome: Change in MMRC Scale From Baseline
Description: • Change from baseline in Modified Medical Research Council (MMRC) dyspnea scale The change from baseline in perceived level of dyspnea over the course of 3 months using the participant's self-reported response to the MMRC. Possible scores are 0, 1, 2, 3 and 4 with higher scores representing severe loss of function due to breathing.
Time Frame: Measurements pre-treatment then at 3 months post-treatment
Population: 191 participants answered the MMRC questionnaire at baseline and again at 3-months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 191
Participants
  MMRC Score 0: number analyzed (Participants) | 13
  MMRC Score 0: Baseline | 3
  MMRC Score 0: 3 Month Follow-Up | 10
  MMRC Score 1: number analyzed (Participants) | 57
  MMRC Score 1: Baseline | 26
  MMRC Score 1: 3 Month Follow-Up | 31
  MMRC Score 2: number analyzed (Participants) | 65
  MMRC Score 2: Baseline | 32
  MMRC Score 2: 3 Month Follow-Up | 33
  MMRC Score 3: number analyzed (Participants) | 179
  MMRC Score 3: Baseline | 86
  MMRC Score 3: 3 Month Follow-Up | 93
  MMRC Score 4: number analyzed (Participants) | 68
  MMRC Score 4: Baseline | 44
  MMRC Score 4: 3 Month Follow-Up | 24

3. Primary Outcome: Change in FEV1 From Baseline
Description: •Change from baseline in FEV1 (COPD patients only) as measured by pulmonary function testing/spirometry.
  The change from baseline in FEV1% predicted as measured by pulmonary function testing/spirometry over the course of 3 months.
Time Frame: Measurements pre-treatment and at 3 months post-treatment
Population: 175 participants with COPD had pulmonary function measurements taken at baseline and at 3-months post-treatment.
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 175
percentage of predicted
  FEV1% Predicted at Baseline | 34.2 (18.1)
  FEV1% Predicted 3-Months Post-Treatment | 35.8 (17.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 1 year for each participant.
Arm/Group | Cell Therapy Treated
All-Cause Mortality (participants affected / at risk) | 23/489
Serious Adverse Events (participants affected / at risk) | 0/489
Other Adverse Events (participants affected / at risk) | 0/489

LIMITATIONS AND CAVEATS:
This study was an observational study only with no control (placebo) group and was designed to examine the outcomes of participants following cellular therapy. This study makes no comparison to placebo or any other treatment. Participants incurred the cost of treatment and travel to the treatment center. This study and treatment protocol was approved by Advarra IRB for Human Subjects Protection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03040674/Prot_001.pdf
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03040674/ICF_002.pdf